CLINICAL TRIAL: NCT07381140
Title: Longitudinal Evaluation of Gut Microbiota and Fecal Metabolome Following Roux-en-Y Gastric Bypass: Clinical Implications and Identification of Predictive Biomarkers
Brief Title: Bariatric Surgery and Gut Microbiota Changes Over Time
Acronym: RYGB-MICROGUT
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Domenica Mallardi, Clinical Researcher (Biologist), Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: RC2026-30
Record Dates: First submitted 2026-01-23; First posted 2026-02-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Obese Patients; Obese Patients With Bariatric Surgery; Gut Microbiota; Healthy Participants
Keywords: gut microbiota; stool metabolome; obesity; bariatric surgery; Roux-en-Y gastric bypass; Long-read sequencing
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This study will collect and retain biological samples to analyze changes in gut microbiota and metabolites in adults undergoing bariatric surgery. The following types of samples will be collected:
  Stool samples - collected at multiple time points before and after RYGB surgery to analyze gut bacterial composition and fecal metabolome.
  Blood samples - collected at the same time points to assess metabolic, inflammatory, and clinical biomarkers.
  Urine samples - collected for additional metabolic analyses and to complement stool and blood data.
  ll samples will be properly labeled, stored, and retained in accordance with applicable institutional and regulatory guidelines. Samples may be used for bacterial DNA-based sequencing analyses, metabolomic profiling, and other related laboratory assays to investigate the relationships between microbiota, metabolites, and clinical outcomes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RYGB Group: Adults aged 18-65 years with severe obesity (BMI ≥ 35 kg/m² with comorbidities or BMI ≥ 40 kg/m²) who are undergoing Roux-en-Y gastric bypass (RYGB) surgery.
- Obese Control Group: Adults aged 18-65 years with obesity (BMI ≥ 30 kg/m²) who are receiving structured dietary treatment without surgery.
- Healthy Control Group: Adults aged 18-65 years with normal weight (BMI 18.5-24.9 kg/m²) and normal metabolic function. This group helps identify normal variations in gut bacteria and metabolites over time, independent of obesity or surgery.

SUMMARY:
The goal of this observational study is to learn how bariatric surgery affects gut bacteria and gut-related metabolic products over time in adults with obesity. The study includes adults aged 18 to 65 years who are undergoing Roux-en-Y gastric bypass (RYGB) surgery, as well as adults with obesity treated with diet alone and healthy normal-weight adults.

The main questions it aims to answer are:

How does bariatric surgery change the composition and diversity of gut bacteria over time? How are these changes related to weight loss and improvement of obesity-related health conditions?

Researchers will compare people undergoing bariatric surgery with people with obesity treated with diet alone and with healthy normal-weight individuals to see if surgery leads to specific changes in gut bacteria and stool metabolites that are linked to better clinical outcomes.

Participants will:

Provide stool samples at scheduled time points over 12 months Provide blood samples and undergo routine clinical assessments Take part in follow-up visits to monitor weight, metabolic health, and gastrointestinal symptoms

DETAILED DESCRIPTION:
Obesity is a complex and multifactorial condition associated with metabolic, inflammatory, and gastrointestinal alterations. In recent years, the gut microbiota has emerged as a key factor involved in energy balance, metabolic regulation, and systemic inflammation. Alterations in gut microbial composition and function have been consistently observed in individuals with obesity and are thought to contribute to metabolic dysfunction.

Bariatric surgery, particularly Roux-en-Y gastric bypass (RYGB), is one of the most effective treatments for severe obesity and its related comorbidities. Beyond weight loss, this procedure induces profound changes in gastrointestinal anatomy and nutrient flow, which may significantly influence the gut microbiota and the metabolites it produces. However, the timing, persistence, and clinical relevance of these microbial and metabolic changes over the long term are not yet fully understood.

This prospective observational study is designed to evaluate longitudinal changes in gut microbiota composition and fecal metabolome following bariatric surgery and to explore their association with clinical and metabolic outcomes. Participants undergoing bariatric surgery will be followed over a 12-month period and compared with individuals with obesity receiving dietary treatment and with healthy normal-weight individuals. This comparative approach allows the identification of changes specifically related to surgery rather than to weight loss alone or to normal temporal variability.

Gut microbiota will be analyzed using DNA-based sequencing approaches, while fecal metabolites will be assessed to capture functional changes in microbial activity. These biological data will be integrated with clinical and laboratory parameters to explore relationships between gut-related changes and outcomes such as weight loss, metabolic improvement, inflammation, and intestinal barrier function.

By providing a longitudinal and integrated view of gut microbiota and metabolome remodeling after bariatric surgery, this study aims to improve understanding of the biological mechanisms underlying surgical outcomes and to support the identification of potential biomarkers that may help predict individual responses and guide more personalized approaches to obesity management.

ELIGIBILITY:
Inclusion Criteria (RYGB Group):

* Age between 18 and 65 years.
* Adults with a body mass index (BMI) ≥ 35 kg/m² with related comorbidities, or BMI ≥ 40 kg/m², who are candidates for Roux-en-Y gastric bypass (RYGB) surgery only.

Exclusion Criteria (RYGB Group):

* Treatment with antibiotics within the last 3 weeks, or probiotics/prebiotics within the last 4-6 weeks, or systemic corticosteroids within the 8 weeks prior to baseline (T0).
* Participation in dietary regimens or calorie restriction programs in the weeks prior to enrollment.
* Chronic inflammatory bowel diseases (e.g., Crohn's disease, ulcerative colitis), ongoing enteric infections, or active neoplasms.
* Previous organ transplant or ongoing systemic immunosuppressive therapy.
* Pregnancy or breastfeeding.
* Previous major gastrointestinal surgery.
* Chronic alcohol consumption above moderate levels or substance use disorder.

Inclusion Criteria (Obese Control Group):

* Age between 18 and 65 years.
* Adults with BMI ≥ 30 kg/m² who are candidates for structured dietary treatment.

Inclusion Criteria (Healthy Control Group):

* Age between 18 and 65 years.
* Normal weight (BMI between 18.5 and 24.9 kg/m²).
* Normal metabolic function: fasting glucose below threshold, normal ALT/AST, no diagnosis of diabetes or metabolic syndrome.
* No chronic gastrointestinal diseases or conditions that could alter the gut microbiota.

Exclusion Criteria (Obese Control and Healthy Control Group):

* Use of antibiotics within the last 3 weeks or probiotics/prebiotics within the last 4-6 weeks.
* Recent gastrointestinal surgery.
* Pregnancy or breastfeeding.
* Extreme diets or recent dietary changes.
* Recent international travel that could have affected the gut microbiota.
* Medications known to influence the gut microbiota (e.g., PPIs, metformin, steroids).
* Active smoking or excessive alcohol consumption.
* Significant gastrointestinal symptoms (chronic diarrhea or constipation).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese subjects attending the clinical nutrition outpatient clinic of the IRCCS "Saverio de Bellis" - Castellana Grotte (BA).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Long-Term Changes in Gut Microbiota After Bariatric Surgery | from enrollment up to 12 months of follow-up
  Longitudinal changes in the composition and diversity of the gut microbiota (alpha diversity, beta diversity, and relative abundance of key bacterial taxa) in patients undergoing Roux-en-Y gastric bypass (RYGB) surgery, assessed using 16S rRNA gene sequencing (short-read and full-length), compared with the Obese Control and Healthy Control groups.

SECONDARY OUTCOMES:
Comparison of Short- and Long-Read 16S Sequencing | from enrollment up to 12 months of follow-up
  Compare the performance of short-read (V3-V4) and long-read (full-length 16S rRNA) sequencing technologies in terms of taxonomic resolution and biomarker identification.
Fecal Metabolome Changes and Predictive Microbe-Metabolite Signatures After Bariatric Surgery | from enrollment up to 12 months of follow-up
  Assess changes in the fecal metabolome over time after bariatric surgery and Identify microbe-metabolite signatures predictive of clinical response to bariatric surgery.
Association Between Gut Microbiota and Clinical Outcomes | from enrollment up to 12 months of follow-up
  Analyze the association between gut microbiota changes and clinical/metabolic parameters (weight loss, comorbidities, inflammatory and intestinal permeability markers)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis, Castellana Grotte, BA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang T, Li H, Ma S, Cao J, Liao H, Huang Q, Chen W. The newest Oxford Nanopore R10.4.1 full-length 16S rRNA sequencing enables the accurate resolution of species-level microbial community profiling. Appl Environ Microbiol. 2023 Oct 31;89(10):e0060523. doi: 10.1128/aem.00605-23. Epub 2023 Oct 6. PMID 37800969
- [Background] Oehler JB, Wright H, Stark Z, Mallett AJ, Schmitz U. The application of long-read sequencing in clinical settings. Hum Genomics. 2023 Aug 8;17(1):73. doi: 10.1186/s40246-023-00522-3. PMID 37553611
- [Background] Salazar N, Ponce-Alonso M, Garriga M, Sanchez-Carrillo S, Hernandez-Barranco AM, Redruello B, Fernandez M, Botella-Carretero JI, Vega-Pinero B, Galeano J, Zamora J, Ferrer M, de Los Reyes-Gavilan CG, Del Campo R. Fecal Metabolome and Bacterial Composition in Severe Obesity: Impact of Diet and Bariatric Surgery. Gut Microbes. 2022 Jan-Dec;14(1):2106102. doi: 10.1080/19490976.2022.2106102. PMID 35903014
- [Background] Palleja A, Kashani A, Allin KH, Nielsen T, Zhang C, Li Y, Brach T, Liang S, Feng Q, Jorgensen NB, Bojsen-Moller KN, Dirksen C, Burgdorf KS, Holst JJ, Madsbad S, Wang J, Pedersen O, Hansen T, Arumugam M. Roux-en-Y gastric bypass surgery of morbidly obese patients induces swift and persistent changes of the individual gut microbiota. Genome Med. 2016 Jun 15;8(1):67. doi: 10.1186/s13073-016-0312-1. PMID 27306058
- [Background] De Luca M, Shikora S, Eisenberg D, Angrisani L, Parmar C, Alqahtani A, Aminian A, Aarts E, Brown W, Cohen RV, Di Lorenzo N, Faria SL, Goodpaster KPS, Haddad A, Herrera M, Rosenthal R, Himpens J, Iossa A, Kermansaravi M, Kow L, Kurian M, Chiappetta S, LaMasters T, Mahawar K, Merola G, Nimeri A, O'Kane M, Papasavas P, Piatto G, Ponce J, Prager G, Pratt JSA, Rogers AM, Salminen P, Steele KE, Suter M, Tolone S, Vitiello A, Zappa M, Kothari SN. Scientific Evidence for the Updated Guidelines on Indications for Metabolic and Bariatric Surgery (IFSO/ASMBS). Obes Surg. 2024 Nov;34(11):3963-4096. doi: 10.1007/s11695-024-07370-7. Epub 2024 Sep 25. PMID 39320627